CLINICAL TRIAL: NCT03033485
Title: 18F-Labeled Picolinamide PET-CT in the Management of Patients With Melanoma: The Radiation Dosimetry and Diagnostic Applications in Melanoma Patients
Brief Title: 18F-Labeled Picolinamide PET Imaging of Melanoma Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20151230-1
Record Dates: First submitted 2016-12-13; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: Picolinamide; PET/CT; Diagnosis; Melanoma
MeSH Terms: conditions — Melanoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melanoma patients (Experimental): Melanoma patients enrolled for the clinical diagnosis study are performed with both 18F-P3BZA PET/CT and18F-FDG PET/CT scans before surgery.
  Interventions: Radiation: 18F-P3BZA

INTERVENTIONS:
Radiation: 18F-P3BZA — 18F-P3BZA is a type of 18F labeled Picolinamide targeting melanin which is highly secreted in Melanoma. The toxicity of P3BZA was evaluated by SoBran Bioscience. The final report showed that there no signs of toxicity during the conduct of the toxicity study. No treatment-related differences were noted in mean body weight and body weight changes, clinical chemistry, haematology, or coagulation parameter after a single intravenous dose of P3BZA at 0.0589mg/kg.
  Other Names: 18F labeled Picolinamide

SUMMARY:
The purpose of this study is to assess the dosimetric properties of the positron emission tomography (PET) imaging probe 18F labeled Picolinamide (18F-P3BZA) and preliminarily evaluate its diagnosis value in melanoma patients.

DETAILED DESCRIPTION:
50 patients with pathology diagnosed melanoma will be enrolled for the clinical study. If agree to take part in this study, the patient will be performed with 18F-P3BZA PET/CT scan and 18F-FDG PET/CT scan in the other day before and after surgery. Next, all of the resected tissues from the patients will be checked with pathology.

6 of 50 patients are performed for whole-body PET scans at 0, 15, 30, 45, 60, and 120 minutes and a CT scan at 60 minutes after tracer injection (mean dose, 5.0 ± 0.5 mCi in 2.0 ± 0.5ml) will be performed. During the imaging period, 1 mL blood samples will be obtained for time-activity curve calculations at 1, 5, 10, 30,60, 90, 120, and 180 minutes after injection. The estimated radiation doses will be calculated by using OLINDA/EXM software.

The images produced by these scans will be compared to see the diagnosis value of 18F-P3BZA.

Screening Tests:

Women who decide to take part in this study will be asked if they think they might be pregnant at the start of the study. All of them must have a negative blood pregnancy test (Human chorionic gonadotropin, HCG).

PET-CT Scan Procedure:

Before the PET-CT scan is performed, patient will be asked to remove any metallic objects when she/he arrive at the PET-CT Center. After a property rest, he/she will be injected with about 5mCi 18F-P3BZA. The first scan will take at 60 minutes after injection and a delay scan will take at 120 minutes after injection. Each PET/CT scan will take about 20 minutes.

After 18F-P3BZA scan, the patient will be asked to avoid stressful exercise. Starting about 12 hours before 18F-FDG scan, he/she will be asked to limit the amount of carbohydrates until the scans are done.

Follow-Up Visits:

Patients' primary care physician will follow-up them for next 24 hours. After then, they may order additional imaging or surgical results after this study for follow-up purposes. The study doctor will review these results to compare them with the PET-CT images. The study doctors will also review the results of any biopsies you may have had as a result of PET-CT findings.

This is an investigational study. PET-CT and CT scans are FDA approved and commercially available.

ELIGIBILITY:
Inclusion Criteria:

* patients with melanoma: diagnosed by pathology and ready for surgery

Exclusion Criteria:

* patients with melanoma: refuse or cannot endure surgery
* pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
SUV of organs and melanoma | 1 hour after injection
  The maximum standardized uptake values (SUVmax) with unit of g/mL of 18F-P3BZA and 18F-FDG in melanoma tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital Nuclear Medicine Department, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No